CLINICAL TRIAL: NCT04332068
Title: A Randomised, Double-blind, Placebo-controlled Trial to Assess the Safety, Pharmacokinetics, and Efficacy of Escalating Doses of Oral Ivermectin in Scabies Infected Children Weighing 5 to Less Than 15 Kilograms
Brief Title: Ivermectin Safety in Small Children
Acronym: ISSC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Fundação Alfredo da Matta (FUAM) (Unknown); Kenya Medical Research Institute (Other); Fundação de Medicina Tropical Doutor Heitor Vieira Dourado (FMT-HVD) (Unknown); Medical Research Center Unit The Gambia (MRCG) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PAR20001
Record Dates: First submitted 2020-03-16; First posted 2020-04-02 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Scabies
Keywords: Scabies; Ivermectin; permethrin
MeSH Terms: conditions — Scabies | interventions — Ivermectin

STUDY DESIGN:
Intervention Model Description: The trial will initially randomize 30 participants at each site to receive control (permethrin cream), ivermectin 200 or 400 µg/kg (10:10:10) and review this data before escalation to ivermectin 800 µg/kg. Once the initial 30 participants have been treated a DSMB consultation will be performed for each site. If deemed safe to escalate to ivermectin 800 µg/kg, then remaining participants at each site will be treated with control (permethrin cream), ivermectin 200, 400, or 800 µg/kg (15: 15: 15: 25).
  The Brazil site will initially randomize 30 participants receive control (permethrin cream) or ivermectin 200 µg/kg (15:15) and review this data before escalation to ivermectin 400 µg/kg. Once the initial 30 participants have been treated a DSMB consultation will be performed. If deemed safe to escalate to ivermectin 400 µg/kg, then remaining participants at the site will be treated with control (permethrin cream), ivermectin 200 or 400 µg/kg (18: 18: 33).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial so the participants, their parents, guardians or carers, administering clinicians, attending nurses, the central research team, and independent outcome assessors will all be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Active Comparator): Permethrin cream plus placebo tablets
  Interventions: Drug: Permethrin Cream; Other: Placebo tablet
- Arm 2 (Experimental): Ivermectin (200 µg/kg) plus placebo cream
  Interventions: Drug: Oral ivermectin; Other: Placebo cream
- Arm 3 (Experimental): Ivermectin (400 µg/kg) plus placebo cream
  Interventions: Drug: Oral ivermectin; Other: Placebo cream
- Arm 4 (Experimental): Ivermectin (800 µg/kg) plus placebo cream (Kenya and The Gambia sites)
  Interventions: Drug: Oral ivermectin; Other: Placebo cream

INTERVENTIONS:
Drug: Oral ivermectin — Ivermectin (NT007) 3 mg tablets are round, white, and scored on one side. Ivermentin 3mg tablets will be crushed and mixed thoroughly in 10mL of water.
  Other Names: NT007, Liconsa Laboratorios
  Arms: Arm 2; Arm 3; Arm 4
Drug: Permethrin Cream — permethrin cream 5% (Pioletal® Plus) is a white coloured lotion with a homogenous appearance and an odour of fennel and lavender.
  Other Names: Pioletal® Plus
  Arms: Arm 1
Other: Placebo tablet — placebo tablets are round, white, scored on one side. There are no active substances in the placebo tablets.
  Arms: Arm 1
Other: Placebo cream — A placebo cream is a white coloured lotion with a homogenous appearance and an odour of fennel and lavender but lacking the permethrin agent.
  Arms: Arm 2; Arm 3; Arm 4

SUMMARY:
This trial will evaluate the safety, pharmacokinetics, and efficacy of ivermectin in scabies infected children weighing 5 to less than 15kg. This will allow future efforts to expand the indication of ivermectin treatment to infants weighing 5 to less than 15kg to treat numerous NTDs, allowing this young age group equitable access to the numerous benefits of ivermectin therapy.

DETAILED DESCRIPTION:
Scabies is a skin infestation caused by a mite called Sarcoptes scabiei. Scabies is characterised by a rash and severe itching, which is an allergic reaction to the eggs and feces the females deposit as they tunnel under the skin. Oral ivermectin is a very safe and beneficial drug which has been shown to be highly effective for the treatment of scabies and more than a dozen different neglected tropical diseases (NTDs), many of which are associated with important public health problems. Current label indications for ivermectin prevent use in small children weighing less than 15 kg, due to limited safety data in this group. Many of the NTD treatment options for small children rely on compounds that are less safe and/or efficacious compared to oral ivermectin. Our proposal will establish the safety and pharmacokinetics of escalating doses of ivermectin (200, 400, 800 µg/kg) to treat scabies infected children weighing 5 to less than 15 kg. The safety assessment will provide crucial evidence on the use of ivermectin for numerous diseases in children weighing 5 to less than 15 kg. The information from measuring drug concentrations in the patients will inform the optimal dosing of this drug in small children. Assessment of the efficacy of ivermectin, compared to permethrin cream, for the treatment of scabies in small children can provide an important alternative treatment for this widespread disease. This trial has been funded by the Wellcome Trust (grant reference number: 218524/Z/19/Z).

ELIGIBILITY:
Inclusion Criteria:

* Male or female child weighing 5 to <15 kilograms
* ≥2 months old
* Scabies infestation
* Available to attend all study visits
* Parents/guardians/carers able to provide consent

Exclusion Criteria:

The participant may not enter the trial if ANY of the following apply:

* A history of renal or hepatic impairment.
* Any other significant disease or disorder (e.g. moderate or severe malnutrition) which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.
* Participants who have participated in another research trial involving an investigational product in the past 12 weeks.
* Children with Crusted/Norwegian scabies or severe secondary bacterial infections (e.g. sepsis)
* Children who have taken ivermectin or topical permethrin cream within the last two weeks
* Children with known allergies to ivermectin or topical permethrin cream or excipients
* Loa loa infection risk, assessed based on travel history to endemic areas
* Use of prescription (especially CYP3A4 inhibitors or inducers) or non-prescription drugs (except paracetamol at doses of up to 90 milligrams/kg/day), including vitamins (especially vitamin C), herbal and dietary supplements (including St. John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 times the drug half-life (whichever is longer) prior to the first dose of study medication until the completion of the follow-up procedure, unless in the opinion of investigator, the medication will not interfere with the study procedures or compromise patient safety; the investigator will take advice from the manufacturer representative as necessary.
* The investigator, health care provider or study staff feel that the patient is not suitable for study participation due to chronic illness, suspected underlying illness, or concerns that the patient will adhere to follow-up schedule.
* Previously treated in the ISSC study

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 240 (Actual)
Dates: Start 2023-11-18 (Actual); Primary Completion 2025-04-04 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Comparing the occurrence of adverse events between the intervention (ivermectin) and control (permethrin) groups | 15 days
  Pruritus will be assessed through physical examination and via diary cards provided to the parents/carers.

SECONDARY OUTCOMES:
Population pharmacokinetic properties of ivermectin at escalating doses | 15 days
  Time to peak plasma concentration (Tmax; hours)
Population pharmacokinetic properties of ivermectin at escalating doses | 15 days
  Peak plasma concentration (Cmax; mg/L)
Population pharmacokinetic properties of ivermectin at escalating doses | 15 days
  Area under the plasma drug concentration-time curve (AUC0-24; mg×h×L-1)
Efficacy of oral ivermectin | 15 days
  Comparing the reduction of dermatological manifestations by "performing physical examination to quantify the number and size of scabies lesions on days 0, 7 and 14" in the oral intervention (oral ivermectin) and control (permethrin cream) groups.

OTHER OUTCOMES:
Pharmacogenomics of ivermectin | day 0
  Whole genome sequencing will be used to determine associations between pharmacogenetic variants with pharmacokinetic or pharmacodynamic parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz von Seidlein, Ass.Prof., Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (3):
- Alfredo da Matta Tropical Dermatology Foundation (FUAM), Manaus, Brazil
- Kenya Medical Research Institute, Kisumu, Kenya
- MRC Unit The Gambia, Banjul, The Gambia

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be under the custodianship of MORU. With participant's consent, data from this study may be shared in a de-identified form with other groups or researchers in accordance with the MORU Data Sharing Policy.
Time Frame: After completion of trial activities and reporting
Access Criteria: MORU Data Sharing Policy. (http://www.tropmedres.ac/data-sharing-policy)